CLINICAL TRIAL: NCT00668200
Title: Post US Approval Voluntary Registry Study to Determine Incidence of Hypocalcemia Post Reclast® Treatment in Patients With Paget's Disease After Institution of Educational Strategies to Improve Adherence to Calcium and Vitamin D Supplementation
Brief Title: Impact on Reducing the Incidence of Low Serum Calcium by Providing Educational Materials on the Need to Take Daily Supplemental Calcium and Vitamin D to Patients With Paget's Disease Treated With Reclast®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446K2401
Record Dates: First submitted 2008-04-22; First posted 2008-04-29 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Paget's Disease of the Bone; Hypocalcemia
Keywords: Paget's; hypocalcemia; zoledronic acid; serum calcium
MeSH Terms: conditions — Osteitis Deformans; Hypocalcemia | interventions — Zoledronic Acid; Calcium; Vitamin D

ARMS (1):
- zoledronic acid (Other): 5 mg of Reclast (ZOL446, zoledronic acid) injection in 100 mL ready to infuse solution administered intravenously via a vented line. The infusion time was to be not less than 15 minutes given over a constant infusion rate.
  Interventions: Drug: Reclast (ZOL446, zoledronic acid); Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Reclast (ZOL446, zoledronic acid) — 5 mg i.v. annually ("real-life, physician prescribed")
  Other Names: Reclast, ZOL446
Dietary Supplement: Calcium — 1500 mg elemental calcium daily in divided doses (the divided doses were 2-3 times per day depending on the formulation)
Dietary Supplement: Vitamin D — 800 IU vitamin D daily, particularly in the immediate 2 weeks following zoledronic acid administration

SUMMARY:
This study will evaluate the impact of investigator and patient education and educational materials to foster calcium and vitamin D supplementation to mitigate the potential for hypocalcemia post Reclast® administration in patients with Paget's disease of bone.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* As per currently approved Reclast® Package Insert:

Exclusion Criteria:

- As per currently approved Reclast® Package Insert:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (9):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Gainesville, Georgia
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Waco, Texas
  - Novartis Investigative Site, Madison, Wisconsin

REFERENCES:
- See also: Related Info — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid
Started | 80
Safety Population | 81 (1 patient was not included in the ITT patient was enrolled in error)
Intent to Treat (ITT) | 80
Completed | 77
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The ITT population includes 80 enrolled patients and the Safety population includes 81enrolled patients. During monitoring it was discovered that one patient signed the consent form from another Paget's study; therefore, this patient was excluded from the ITT population but included in the safety population.Baseline used ITT data set
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (12.98) [39 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Serum Calcium <2.07 mmol/L at 9-11 Days After Receiving Zoledronic Acid.
Description: To be included in the analysis, patients were required to have a baseline serum calcium of at least 2.07 mmol/L and at least one serum calcium measurement 9-11 days post-infusion of zoledronic acid. In case of multiple assessments, for baseline visit the last measurement prior to the first dose was used in the analysis, and for Visits 2 and 3, the lowest serum calcium in the visit window was used. hypocalcemia was defined as treatment-emergent serum calcium <2.07 mmol/L at 9-11 days after the study drug infusion.
Time Frame: at Visit 2 (days 9 - 11 post-infusion), visit 3 (day 30)
Population: Safety population which includes 81 patients was used. 75 of the 81 patients in the safety population met the criteria. 6 patients did not meet criteria and were excluded from the analysis: 1 patient had a low serum calcium at baseline, and the other 5 patients were missing serum calcium values either at baseline or post-baseline.
Measure: Number; unit: percentage of patients
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 75
percentage of patients
  Visit 2 | 1.3
  Visit 3 | 0.0

2. Secondary Outcome: Change From Baseline in Serum Calcium (mmol/L) - Safety Population
Description: Change from baseline = endpoint - baseline, at each time point, only participants with a value at baseline and that time point are included in the change from baseline column. In case of multiple assessments, for baseline visit the last measurement prior to the first dose was used in the analysis, and for Visits 2 and 3, the lowest serum calcium in the visit window was used.
Time Frame: Baseline, Visit 2 (days 9 - 11 post-infusion), visit 3 (day 30)
Population: This Outcome Measure uses Safety population which includes 81 patients. During monitoring it was discovered that one patient signed the consent form from another Paget's study; therefore, this patient was excluded from the ITT population but included in the safety. The ITT population was used for participant flow and baseline characteristics.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 81
mmol/L
  Visit 2 n=76 | -0.024 (0.189)
  Visit 3 n=2 | 0.04 (0.014)

3. Secondary Outcome: Percentage of Newly Occurring Post-baseline Hypocalcemia Symptoms Based on Hypocalcemia Questionnaire at End of Study Visit 2 or Visit 3 (Safety Population)
Description: The end of study is not a separate time point. It is the last post-baseline, for majority the end of study was visit 2. There were 2 patients who had the end of study at Visit 3. If calcium at visit 2 was abnormal it was measured again at visit 3.
Time Frame: End of study: Visit 2 (days 9 - 11 post-infusion) or visit 3 (day 30)
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 81
percentage of patients
  Tingling around your mouth n=76 | 1.3
  Tingling in fingers n=66 | 3
  Cramps in hands n=62 | 3.2
  Cramps in leg or feet n=50 | 0
  Involuntary movements of hands n=73 | 2.7
  Involuntary movements of feet n=70 | 1.4
  Involuntary movements of facial muscles n=71 | 0
  Generalized (epileptic) seizures n=76 | 0

ADVERSE EVENTS:
Arm/Group | Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 1/81
Other Adverse Events (participants affected / at risk) | 24/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=81)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=81)
Acute phase reaction (General disorders) | 6
Chills (General disorders) | 10
Malaise (General disorders) | 6
Pain (General disorders) | 9
Pyrexia (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.